CLINICAL TRIAL: NCT04652752
Title: A Prospective, Open, Clinical Trial to Evaluate the Safety and Efficacy of Dressing CONNETTIVINA HI TECH in the Management of Superficial Cutaneous Lesions
Brief Title: Clinical Investigation to Evaluate the Safety and Efficacy of Dressing CONNETTIVINA HI TECH in the Management of Superficial Cutaneous Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment Difficulties
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AQ04-19-01
Record Dates: First submitted 2020-03-02; First posted 2020-12-03 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Superficial Cutaneous Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONNETTIVINA HI TECH patch (Experimental): CONNETTIVINA HI TECH patch will be applied to eligible patients. CONNETTIVINA HI TECH will be renewed every two day, according with general principles of wound management
  Interventions: Device: CONNETTIVINA HI TECH patch

INTERVENTIONS:
Device: CONNETTIVINA HI TECH patch — It is a medical device for topical application in the form of a patch with adhesive transparent polyurethane edge and a central pad impregnated with a solution of hyaluronic acid sodium salt, able to create a hydrating environment, such as to favor the natural healing process of tissue repair in case of bruises, abrasions, small cuts, superficial wounds, burns

SUMMARY:
This is an open, single arm, prospective clinical investigation to evaluate the performance of CONNETTIVINA HI TECH, in terms of safety and efficacy in the management of superficial cutaneous lesions. The study will be conducted in one center, in Italy and will enroll 50 subjects . Subjects will be followed until confirmation of complete wound closure, and for a maximum of 26 days, with a follow up of 4 days after re-epithelization will be confirmed.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Male or female ≥ 18 and ≤ 85 years
* Having a superficial cutaneous lesion of different etiology, with the following characteristics:

Wound bed appearance of grade ≥15 of WBS (Wound Bed Score: Falanga 2006) Absence of clinical signs or symptoms of local infection (as defined by CDC/NHSN) Size: between 5 and 32 cm2 that can be covered by a dressing of 4x8cm

* In case of multiple lesions per patient, only one lesion will be considered for the treatment (the better choice for self-evaluation of lesion by patient)
* Patient able to maintain a Patient's Diary during the study
* Patient able to read and understand the language and content of the study material, understand the requirements for follow-up visits, is willing to provide information at the scheduled evaluations and is willing and able to comply with the study requirements
* Ensured compliance of subjects for the study period

Exclusion Criteria:

1. Patients who not sign the informed consent form
2. Patients with non-superficial wounds exposing bones, tendon or muscle bundles.
3. Patients with WBS score under or equal to 14 ("severe exudate amount", or "moderate exudate amount" and "moderate per-wound dermatitis" or "moderate callous peri-wound")
4. Presence of signs of infection as defined by CDC/NHMS
5. History of connective tissue disease, e.g., systemic lupus erythematosus, systemic sclerosis, Sjögren's syndrome or mixed connective tissue disease
6. Uncontrolled congestive heart failure
7. Active malignant disease
8. Active sickle cell disease
9. Patients who are immunocompromised for reasons such as therapy with corticosteroids, chemotherapy, antiangiogenic or immunosuppressive agents, or due to immunodeficiency syndromes
10. Known allergy to any of the devices' constituents
11. Women who are pregnant, breastfeeding or who have not reached menopause and are not abstinent or practicing an acceptable means of birth control as determined by the Investigator for the duration of the study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in dimentions of lesion in patients compared to baseline | at 14 days
  Change from of superficial cutaneous lesions by measuring the area of the superficial lesion after 14 days of treatment

SECONDARY OUTCOMES:
Healing rate as a difference in the mean percentage reduction of lesion area from baseline in patients treated with CONNETTIVINA HI TECH | at 2,8, 14, 20 and 26 days
  The healing rate will be evaluated at all time points as a difference in the mean percentage reduction of lesion area from baseline measured by a wound imaging device
Patient's satisfaction with CONNETTIVINA HI TECH | at 2,8, 14, 20 and 26 days
  Patient's satisfaction with CONNETTIVINA HI TECH will be evaluated at each post baseline visit: patients will assess their degrees of satisfaction with the use of the dressing by the means of a 5 grade scale
Clinician's global assessment of the lesion (CGA) | at 2,8, 14, 20 and 26 days
  Clinical Global Assessment (CGA) will be evaluated at each post baseline visit: the clinician will be requested to score the lesion on a five grade scale
Evaluation of dressing Adhesion | at day 28
  Evaluation of dressing adhesion evaluated at each visit by considering the effective frequency of dressing change and comparing it with the frequency indicated by the clinical investigation plan
Number of Participants With Treatment-Related Adverse Events | at 2,8, 14, 20 and 26 days
  The safety and tolerability of treatments will be assessed by investigating local and expected adverse events, as consequence of the product application and any other adverse event occurred during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Iperbarico di Ravenna, Ravenna, Italy